CLINICAL TRIAL: NCT06989684
Title: Implant Stability And Changes In Ridge Width Using Underdrilling Versus Osseodensification Protocols For Posterior Dental Implant- A Randomized Clinical Trial
Brief Title: Implant Stability Changes Using Underdrilling Versus Osseodensification Protocols for Posterior Dental Implants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHAINSHILPA-PERIO
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Dental Implant Stability
Keywords: secondary implant stability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blinding will be performed. The patient, the outcome assessor and data analyst will be blinded to the allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Osseodensification (Active Comparator): Osseodensification uses special densa burs for osteotomy site compaction
  Interventions: Procedure: Osseodensification
- Underilling (Active Comparator): In Underdrilling the osteotomy is smaller than implant diameter to be placed
  Interventions: Procedure: Underdrilling

INTERVENTIONS:
Procedure: Osseodensification — Osseodensification uses specially designed burs to densify osteotomy site
  Arms: Osseodensification
Procedure: Underdrilling — In underdrilling the osteotomy is smaller than implant diameter to be placed
  Arms: Underilling

SUMMARY:
This clinical trial aims to compare two drilling protocols Underdrilling and Osseodensification for placing dental implants in patients with low bone density. The purpose is to compare which technique provides better primary and secondary implant stability in the posterior regions of the jaw with low bone density. The hypothesis is that there is no significant difference in implant stability between the two protocols.

DETAILED DESCRIPTION:
Achieving sufficient primary stability becomes difficult in areas with low bone density. One technique commonly used is Underdrilling protocol.With the Underdrilling technique, the final osteotomy is smaller than the diameter of the implant to be placed.A relatively new Osseodensification protocol, introduced by Huwais in 2013, employs specially designed bur that smoothly compact the bone as they expand an osteotomy. This may prove to be particularly helpful in cases with low bone quality.This clinical trial aims to compare the implant stability using these drilling protocols

ELIGIBILITY:
Inclusion Criteria:

1. Patient partially edentulous ridge after extraction of more than 6 months and with low bone density.
2. Systemically healthy patients ≥18 years of age.

Exclusion Criteria:

1. Smokers.
2. Pregnant or lactating females.
3. Uncontrolled systemic disease like diabetes, hypertension, hormonal therapy and hematologic diseases.
4. History of Maxillary sinus pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 12-18 months
  It compares Primary stability and Secondary stability after implant placement. Primary stability is recorded by insertion torque values from manual torque wrench. Secondary stability is recorded by resonance frequency analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Ritika Arora, MDS, Principal Investigator — PGIDS,Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No